CLINICAL TRIAL: NCT00252941
Title: The Role Of Prophylactic Urethral Stenting With Memokath® 028SW in Patients Undergoing Prostate 125I Seed Implants For Prostate Carcinoma: A Phase I/II Study
Brief Title: Prophylactic Urethral Stenting With Memokath After Prostate Implantation for Prostate Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 8488; CASE16804
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Prostate Cancer; Post-Brachytherapy Bladder Outlet Obstruction
Keywords: prostate cancer; brachytherapy; urethral stenting
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Device: Memokath 028SW Urethral Stent

SUMMARY:
The purpose of this study is to determine the feasibility, safety, and efficacy of the Memokath® 028SW stent to prevent urinary obstructive symptoms (difficulty urinating) when used after prostate seed implantation for the treatment of localized prostate cancer.

DETAILED DESCRIPTION:
Image-guided transperineal permanent prostate brachytherapy (PI) is an accepted curative treatment option for patients with early stage prostate cancer. Multiple reports have defined its efficacy and shown it to be superior to antecedent trans-abdominal techniques. In addition, the efficacy of PI has been shown to be similar to radical retropubic prostatectomy (RRP) and external beam radiotherapy (EBRT). These positive results, however, are gained at the expense of toxicity. The most notable toxicity is associated with the urinary system. The most severe side effect of PI is urinary retention requiring intermittent self-catheterization (ISC).

The reported rate of severe urinary retention following PI is ~10%. Most of these patients can be managed with ISC and alpha-blockers for a few weeks. Although this is generally a temporary phenomenon, a small percentage will eventually require surgical intervention to permit urinary flow. This is a major concern for patients undergoing PI, but should not be a reason to avoid this form of curative treatment.

The use of implantable stents has been successful in BPH. The Memokath® device has been shown to decrease the International Prostate Symptom Score from a mean of 20.3 to 8.2 in the first 3 months after stent placement in patients with bladder outlet obstruction unable to undergo TURP. Few experience side-effects with pain in 3%, hematuria in 3%, incontinence in 6%, and infection in 6%. A multicenter randomized control trial is currently underway assessing the use of this device in patients with recurrent urethral strictures.

Urethral stents have been used with some success in patients with post-brachytherapy bladder outlet obstruction. Five patients, who could not tolerate alpha-blockers or clean intermittent catheterization, received UroLume urethral stents following one or more episodes of urinary retention. All patients were able to void immediately after stent placement. No patients developed incontinence after the stent placement. The main complaints following UroLume® stent placement were urethral bleeding, referred pain at the head of the penis, and dysuria. These symptoms required stent removal in 2 out of the 5 patients. In another study, five patients received SpannerTM urethral stents following significant urinary symptoms after prostate brachytherapy. All patients were able to void spontaneously with no post-void residual volume of urine. Flow rates increased and the International Prostate Symptom Score decreased from a mean of 25.2 to 10 (p=0.03). However, two patients experienced pain, which required removal of the stent.

Given that few patients have experienced side effects with the Memokath® urethral stent in bladder outlet obstruction, we wish to assess the toxicity associated with this stent in a post-brachytherapy setting. In addition, we would like to assess its efficacy when used prophylactically in reducing bladder outlet obstruction following prostate brachytherapy and its impact on the AUA score.

ELIGIBILITY:
Inclusion Criteria:

* eligible for prostate seed implant
* 50 years of age or older
* able to give informed consent

Exclusion Criteria:

* presence of any other urologic implant, including stents,penile prosthesis or artificial sphincter
* history of transurethral resection of prostate (TURP)procedure
* presence of urethral diverticuli
* presence of urethral strictures
* presence of bladder calculi or tumors
* prostatic urethra is less than 2.5 cm or greater than 6.5 cm
* inability to participate in study activities due to physical or mental limitations
* inability or unwillingness to return for all the required follow-up visits

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-11; Primary Completion 2006-04 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Morbidities assessed on RTOG Morbidity Scale weekly for 12 weeks after PI then biweekly for next 12 weeks
Clinic visits at 2 weeks, 3 months and 6 months; physical exam to include urine flow rate, post-void residual and urinalysis
CT at 1 month post-brachytherapy
Device removal at 6 months (earlier if adverse event or patient wishes to discontinue trial)
Cystoscopy to assess urethra after stent removal

SECONDARY OUTCOMES:
AUA score to assess severity of urinary symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jay P Ciezki, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Ragde H, Blasko JC, Grimm PD, Kenny GM, Sylvester JE, Hoak DC, Landin K, Cavanagh W. Interstitial iodine-125 radiation without adjuvant therapy in the treatment of clinically localized prostate carcinoma. Cancer. 1997 Aug 1;80(3):442-53. doi: 10.1002/(sici)1097-0142(19970801)80:33.0.co;2-x. PMID 9241078
- [Background] Ragde H, Korb LJ, Elgamal AA, Grado GL, Nadir BS. Modern prostate brachytherapy. Prostate specific antigen results in 219 patients with up to 12 years of observed follow-up. Cancer. 2000 Jul 1;89(1):135-41. PMID 10897010
- [Background] Blasko JC, Ragde H, Grimm PD. Transperineal ultrasound-guided implantation of the prostate: morbidity and complications. Scand J Urol Nephrol Suppl. 1991;137:113-8. PMID 1947828
- [Background] Kleinberg L, Wallner K, Roy J, Zelefsky M, Arterbery VE, Fuks Z, Harrison L. Treatment-related symptoms during the first year following transperineal 125I prostate implantation. Int J Radiat Oncol Biol Phys. 1994 Mar 1;28(4):985-90. doi: 10.1016/0360-3016(94)90119-8. PMID 8138452
- [Background] Terk MD, Stock RG, Stone NN. Identification of patients at increased risk for prolonged urinary retention following radioactive seed implantation of the prostate. J Urol. 1998 Oct;160(4):1379-82. PMID 9751358
- [Background] Benoit RM, Naslund MJ, Cohen JK. A comparison of complications between ultrasound-guided prostate brachytherapy and open prostate brachytherapy. Int J Radiat Oncol Biol Phys. 2000 Jul 1;47(4):909-13. doi: 10.1016/s0360-3016(00)00506-x. PMID 10863059
- [Background] Lee N, Wuu CS, Brody R, Laguna JL, Katz AE, Bagiella E, Ennis RD. Factors predicting for postimplantation urinary retention after permanent prostate brachytherapy. Int J Radiat Oncol Biol Phys. 2000 Dec 1;48(5):1457-60. doi: 10.1016/s0360-3016(00)00784-7. PMID 11121648
- [Background] Bruno JF, Whittaker J, Song JF, Berelowitz M. Molecular cloning and sequencing of a cDNA encoding a human alpha 1A adrenergic receptor. Biochem Biophys Res Commun. 1991 Sep 30;179(3):1485-90. doi: 10.1016/0006-291x(91)91740-4. PMID 1656955
- [Background] Ramarao CS, Denker JM, Perez DM, Gaivin RJ, Riek RP, Graham RM. Genomic organization and expression of the human alpha 1B-adrenergic receptor. J Biol Chem. 1992 Oct 25;267(30):21936-45. PMID 1328250
- [Background] Lepor H. Phase III multicenter placebo-controlled study of tamsulosin in benign prostatic hyperplasia. Tamsulosin Investigator Group. Urology. 1998 Jun;51(6):892-900. doi: 10.1016/s0090-4295(98)00126-5. PMID 9609623
- [Background] Lepor H. Long-term evaluation of tamsulosin in benign prostatic hyperplasia: placebo-controlled, double-blind extension of phase III trial. Tamsulosin Investigator Group. Urology. 1998 Jun;51(6):901-6. doi: 10.1016/s0090-4295(98)00127-7. PMID 9609624
- [Background] Chapple CR, Wyndaele JJ, Nordling J, Boeminghaus F, Ypma AF, Abrams P. Tamsulosin, the first prostate-selective alpha 1A-adrenoceptor antagonist. A meta-analysis of two randomized, placebo-controlled, multicentre studies in patients with benign prostatic obstruction (symptomatic BPH). European Tamsulosin Study Group. Eur Urol. 1996;29(2):155-67. PMID 8647141
- [Background] Schulman CC, Cortvriend J, Jonas U, Lock TM, Vaage S, Speakman MJ. Tamsulosin, the first prostate-selective alpha 1A-adrenoceptor antagonist. Analysis of a multinational, multicentre, open-label study assessing the long-term efficacy and safety in patients with benign prostatic obstruction (symptomatic BPH). European Tamsulosin Study Group. Eur Urol. 1996;29(2):145-54. PMID 8647140
- [Background] Elshaikh MA, Ulchaker JC, Reddy CA, Angermeier KW, Klein EA, Chehade N, Altman A, Ciezki JP. Prophylactic tamsulosin (Flomax) in patients undergoing prostate 125I brachytherapy for prostate carcinoma: final report of a double-blind placebo-controlled randomized study. Int J Radiat Oncol Biol Phys. 2005 May 1;62(1):164-9. doi: 10.1016/j.ijrobp.2004.09.036. PMID 15850917
- [Background] Perry MJ, Roodhouse AJ, Gidlow AB, Spicer TG, Ellis BW. Thermo-expandable intraprostatic stents in bladder outlet obstruction: an 8-year study. BJU Int. 2002 Aug;90(3):216-23. doi: 10.1046/j.1464-410x.2002.02888.x. PMID 12133055
- [Background] Konety BR, Phelan MW, O'Donnell WF, Antiles L, Chancellor MB. Urolume stent placement for the treatment of postbrachytherapy bladder outlet obstruction. Urology. 2000 May;55(5):721-4. doi: 10.1016/s0090-4295(00)00486-6. PMID 10792088
- [Background] Henderson A, Laing RW, Langley SE. A Spanner in the works: the use of a new temporary urethral stent to relieve bladder outflow obstruction after prostate brachytherapy. Brachytherapy. 2002;1(4):211-8. doi: 10.1016/S1538-4721(02)00100-9. PMID 15062169
- [Background] Nag S, Beyer D, Friedland J, Grimm P, Nath R. American Brachytherapy Society (ABS) recommendations for transperineal permanent brachytherapy of prostate cancer. Int J Radiat Oncol Biol Phys. 1999 Jul 1;44(4):789-99. doi: 10.1016/s0360-3016(99)00069-3. PMID 10386635
- [Background] Nag S, Bice W, DeWyngaert K, Prestidge B, Stock R, Yu Y. The American Brachytherapy Society recommendations for permanent prostate brachytherapy postimplant dosimetric analysis. Int J Radiat Oncol Biol Phys. 2000 Jan 1;46(1):221-30. doi: 10.1016/s0360-3016(99)00351-x. PMID 10656396